CLINICAL TRIAL: NCT05392153
Title: The Effect of Myofascial Release Technique on Sportive Performance, Balance and Injury Risk in Runners.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2678
Record Dates: First submitted 2022-05-10; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: Runt
Keywords: myofascial release; run; performance; balance; injury risk; fascia
MeSH Terms: conditions — Dwarfism | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial therapy group (Experimental): The myofascial therapy group (n=26) will receive 12 sessions of 6-weekly lower extremity posterior muscle myofascial therapy.
  Interventions: Other: Myofascial therapy
- Control group (No Intervention): The control group (n=23) will not receive lower extremity posterior muscle myofascial therapy. They will continue the routine exercise program.

INTERVENTIONS:
Other: Myofascial therapy — Running is a sport that involves repetitive movement and is particularly vulnerable to injury in the lower extremities. Myofascial release, on the other hand, is a manual method that is effective in increasing blood and oxygen permeability between tissues, renewing the tissue, protecting it from injury and increasing performance. The aim of our study is to investigate the effect of Myofascial therapy on sportive performance balance and injury risk in runners. The study will carry out on runners with a 3-month running history.
  Other Names: Cross-hand technique
  Arms: Myofascial therapy group

SUMMARY:
In order to investigate the effect of myofascial release technique on sportive performance, balance and injury risk in runners, 49 athletes will include in the study. The myofascial application group (n=26)will receive 12 sessions of 6-weekly lower extremity posterior muscle therapy. The control group (n=23) will continue the routine exercise program.

DETAILED DESCRIPTION:
Running is a sport that involves repetitive movement and is particularly vulnerable to injury in the lower extremities. Myofascial release, on the other hand, is a manual method that is effective in increasing blood and oxygen permeability between tissues, renewing the tissue, protecting it from injury and increasing performance. The aim of our study is to investigate the effect of Myofascial application on sportive performance balance and injury risk in runners. The study will carry out on runners with a 3-month running history. Myofascial application group (n=26) and control group (n=23) will divide into two groups as randomized controlled. My Jump 2 App, Y balance test and Functional Movement Analysis (FMS) will use as assessment methods. The myofascial application group will receive 12 sessions of 6 weeks of therapy for the lower extremity posterior group muscles. The control group will continue the routine exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Have a running history of more than 3 months
* Be between 18 and 45 years old
* Being a healthy individual without chronic disease
* No acute injury affecting the lower extremity
* Running at least 5 km a week
* Willingness to participate in the research

Exclusion Criteria:

* Pregnancy or suspected pregnancy
* Use of alcohol or active substance
* Having another ongoing treatment process
* Having a history of surgery on the lower extremity
* Refusal to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The effect of myofascial release technique on sportive performance | Baseline and 6th week
  Vertical jump test (My jump 2 App.) is a valid, reliable, and useful tool for measuring vertical jump in recreationally active adults

SECONDARY OUTCOMES:
The effect of myofascial release technique on balance | Baseline and 6th week
  Y balance test is a functional movement screening device commonly used to predict the risks of injury in athletes.
The effect of myofascial release technique on injury risk | Baseline and 6th week
  The Functional Movement Screen (FMS) was designed to identify functional movement deficits and asymmetries that may be predictive of general musculoskeletal conditions and injuries, with an ultimate goal of being able to modify the identified movement deficits through individualized exercise prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Kutlutürk Yıkılmaz, PhD, Study Chair — Medipol University
Locations (1):
- Backtofit, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hreljac A. Impact and overuse injuries in runners. Med Sci Sports Exerc. 2004 May;36(5):845-9. doi: 10.1249/01.mss.0000126803.66636.dd. PMID 15126720
- [Background] Adstrum S, Hedley G, Schleip R, Stecco C, Yucesoy CA. Defining the fascial system. J Bodyw Mov Ther. 2017 Jan;21(1):173-177. doi: 10.1016/j.jbmt.2016.11.003. Epub 2016 Nov 16. PMID 28167173
- [Background] Sullivan KM, Silvey DB, Button DC, Behm DG. Roller-massager application to the hamstrings increases sit-and-reach range of motion within five to ten seconds without performance impairments. Int J Sports Phys Ther. 2013 Jun;8(3):228-36. PMID 23772339
- [Background] LeBauer A, Brtalik R, Stowe K. The effect of myofascial release (MFR) on an adult with idiopathic scoliosis. J Bodyw Mov Ther. 2008 Oct;12(4):356-63. doi: 10.1016/j.jbmt.2008.03.008. Epub 2008 Jun 4. PMID 19083694
- [Background] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Background] Chaudhry H, Schleip R, Ji Z, Bukiet B, Maney M, Findley T. Three-dimensional mathematical model for deformation of human fasciae in manual therapy. J Am Osteopath Assoc. 2008 Aug;108(8):379-90. doi: 10.7556/jaoa.2008.108.8.379. PMID 18723456
- [Background] Schleip R, Findley TW, Chaitow L, Huijing PA. Review of Fascia: The Tensional Network of the Human Body. 3. Baskı, E-book: Churchill Livingstone, 2012.
- [Background] Emery CA, Cassidy JD, Klassen TP, Rosychuk RJ, Rowe BB. Development of a clinical static and dynamic standing balance measurement tool appropriate for use in adolescents. Phys Ther. 2005 Jun;85(6):502-14. PMID 15921472
- [Background] Shumway-Cook A, Horak FB. Assessing the influence of sensory interaction of balance. Suggestion from the field. Phys Ther. 1986 Oct;66(10):1548-50. doi: 10.1093/ptj/66.10.1548. No abstract available. PMID 3763708
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Robinson RH, Gribble PA. Support for a reduction in the number of trials needed for the star excursion balance test. Arch Phys Med Rehabil. 2008 Feb;89(2):364-70. doi: 10.1016/j.apmr.2007.08.139. PMID 18226664
- [Background] Landis SE, Baker RT, Seegmiller JG. NON-CONTACT ANTERIOR CRUCIATE LIGAMENT AND LOWER EXTREMITY INJURY RISK PREDICTION USING FUNCTIONAL MOVEMENT SCREEN AND KNEE ABDUCTION MOMENT: AN EPIDEMIOLOGICAL OBSERVATION OF FEMALE INTERCOLLEGIATE ATHLETES. Int J Sports Phys Ther. 2018 Dec;13(6):973-984. PMID 30534463
- [Background] Philp F, Blana D, Chadwick EK, Stewart C, Stapleton C, Major K, Pandyan AD. Study of the measurement and predictive validity of the Functional Movement Screen. BMJ Open Sport Exerc Med. 2018 May 7;4(1):e000357. doi: 10.1136/bmjsem-2018-000357. eCollection 2018. PMID 29765700
- [Background] Kraemer WJ, Mazzetti SA, Nindl BC, Gotshalk LA, Volek JS, Bush JA, Marx JO, Dohi K, Gomez AL, Miles M, Fleck SJ, Newton RU, Hakkinen K. Effect of resistance training on women's strength/power and occupational performances. Med Sci Sports Exerc. 2001 Jun;33(6):1011-25. doi: 10.1097/00005768-200106000-00022. PMID 11404668
- [Background] Spiteri T, Binetti M, Scanlan AT, Dalbo VJ, Dolci F, Specos C. Physical Determinants of Division 1 Collegiate Basketball, Women's National Basketball League, and Women's National Basketball Association Athletes: With Reference to Lower-Body Sidedness. J Strength Cond Res. 2019 Jan;33(1):159-166. doi: 10.1519/JSC.0000000000001905. PMID 28368952
- [Background] Janz KF, Letuchy EM, Burns TL, Francis SL, Levy SM. Muscle Power Predicts Adolescent Bone Strength: Iowa Bone Development Study. Med Sci Sports Exerc. 2015 Oct;47(10):2201-6. doi: 10.1249/MSS.0000000000000648. PMID 25751769
- [Background] Yingling VR, Castro DA, Duong JT, Malpartida FJ, Usher JR, O J. The reliability of vertical jump tests between the Vertec and My Jump phone application. PeerJ. 2018 Apr 20;6:e4669. doi: 10.7717/peerj.4669. eCollection 2018. PMID 29692955
- [Background] Gallardo-Fuentes F, Gallardo-Fuentes J, Ramirez-Campillo R, Balsalobre-Fernandez C, Martinez C, Caniuqueo A, Canas R, Banzer W, Loturco I, Nakamura FY, Izquierdo M. Intersession and Intrasession Reliability and Validity of the My Jump App for Measuring Different Jump Actions in Trained Male and Female Athletes. J Strength Cond Res. 2016 Jul;30(7):2049-56. doi: 10.1519/JSC.0000000000001304. PMID 27328276
- [Background] Haynes T, Bishop C, Antrobus M, Brazier J. The validity and reliability of the My Jump 2 app for measuring the reactive strength index and drop jump performance. J Sports Med Phys Fitness. 2019 Feb;59(2):253-258. doi: 10.23736/S0022-4707.18.08195-1. Epub 2018 Mar 27. PMID 29589412
- [Background] Bosco C, Luhtanen P, Komi PV. A simple method for measurement of mechanical power in jumping. Eur J Appl Physiol Occup Physiol. 1983;50(2):273-82. doi: 10.1007/BF00422166. PMID 6681758
- [Background] Markovic G, Dizdar D, Jukic I, Cardinale M. Reliability and factorial validity of squat and countermovement jump tests. J Strength Cond Res. 2004 Aug;18(3):551-5. doi: 10.1519/1533-4287(2004)182.0.CO;2. PMID 15320660